CLINICAL TRIAL: NCT04433247
Title: Pilot Testing Virtual Delivery of the Body Project Eating Disorder Prevention Program
Brief Title: Peer-Led Dissonance Eating Disorder Prevention: Virtual Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Eric Stice, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 54596
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Eating Disorders
Keywords: Prevention; Peer Leader; Feeding and Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor at post-test and 6 month follow-up are blind to participant randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Led Group Intervention (Experimental): In the virtual peer-led group Intervention, participants voluntarily engage in verbal, written, and behavioral exercises in which they critique and discuss the costs of pursuing the thin-ideal ideal. The intervention is 4 sessions long (1-hr each) and is administered by trained peer facilitators who use an intervention script. Participants will be asked to complete weekly home exercises throughout the course of the intervention.
  Interventions: Behavioral: Peer Led Group Intervention
- Wait-List Control (No Intervention): Participants will be placed on a wait list for four weeks, an equal span of time of participants in the peer led group intervention. At four weeks, participants will complete their post-test assessment, then receive the intervention.

INTERVENTIONS:
Behavioral: Peer Led Group Intervention — Four week dissonance-based program wherein women with body image concerns complete verbal, written, and behavioral activities. The program consist of four 60-minute sessions.
  Other Names: Body Project
  Arms: Peer Led Group Intervention

SUMMARY:
This proposed pilot study will evaluate whether this body acceptance class produces greater reductions in eating disorder risk factor symptoms (pursuit of the thin ideal, body dissatisfaction, dieting, dietary restraint and negative affect), eating disorder symptoms, and future onset of eating disorders over 6-month follow-up in this population.

DETAILED DESCRIPTION:
Dozens of eating disorder prevention programs have been evaluated, but only the 4-hr Body Project has reduced eating disorder symptoms and future eating disorder onset over 3-4 year follow-up, produced larger reductions in outcomes than credible alternative interventions, been shown to engage the intervention target (valuation of the thin beauty ideal), and produced effects in trials from several independent teams. Although undergraduate peer-educator-led Body Project groups have produced larger reductions in outcomes than an eating disorder education video, an unmoderated Internet-based prevention program, and even clinician-led Body Project groups, it can be logistically difficult to schedule in-person Body Project groups with high school and college students. One solution to this key implementation barrier is to have peer educators deliver Body Project groups virtually over the Internet. A pilot trial in Sweden provided initial evidence that virtually-delivered peer-led Body Project groups produced greater reductions in eating disorder symptoms and future onset of eating disorders than an active expressive-writing intervention. The proposed pilot study will evaluate whether Body Project produces greater reductions in risk factor symptoms, eating disorder symptoms, and future onset of eating disorders in this population.

Participation in the intervention will last four weeks. Participants will be randomly assigned to the intervention condition or waitlist-control condition. Assessments will take place at pre-intervention, post-intervention, and 6 month follow up. Waitlist control participants will receive the intervention after they complete their post-test assessment.

ELIGIBILITY:
Inclusion Criteria:

* Body image concerns

Exclusion Criteria:

* N/A

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change over time in Body Dissatisfaction | pre intervention obtained on intake, immediately post intervention, and 6-months after the conclusion of the intervention
  Ten items from the Satisfaction and Dissatisfaction with Body Parts Scale assessed satisfaction with body parts with a response scale ranging from 1 = extremely dissatisfied to 6 = extremely satisfied
Change over time in Thin Ideal Internalization | pre intervention obtained on intake, immediately post intervention, and 6-months after the conclusion of the intervention
  The eight-item Ideal-Body Stereotype Scale-Revised will assess endorsement of the thin beauty ideal using a response scale ranging from 1 = strongly disagree to 5 = strongly agree.

SECONDARY OUTCOMES:
Change over time in Negative Affect | pre intervention obtained on intake, immediately post intervention, and 6-months after the conclusion of the intervention
  Twenty items from the sadness, guilt, and fear/anxiety subscales from the Positive Affect and Negative Affect Scale-Revised will assess negative affect. Participants reported the extent to which they had felt negative emotions on scales ranging from 1 = very slightly or not at all to 5 = extremely.
Change over time in Dieting | pre intervention obtained on intake, immediately post intervention, and 6-months after the conclusion of the intervention
  The 10-item Dutch Restrained Eating Scale will assess the frequency of dieting behaviors using a response scale ranging from 1 = never to 5 = always.
Change over time in Eating Disorder symptoms | pre intervention obtained on intake, immediately post intervention, and 6-months after the conclusion of the intervention
  Interviewer assesses frequency of eating disorder behaviors using Eating Disorder Diagnostic Interview

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stice E, Bohon C, Shaw H, Desjardins CD. Efficacy of virtual delivery of a dissonance-based eating disorder prevention program and evaluation of a donation model to support sustained implementation. J Consult Clin Psychol. 2023 Mar;91(3):139-149. doi: 10.1037/ccp0000796. Epub 2023 Feb 6. PMID 36745074